CLINICAL TRIAL: NCT04082624
Title: Workplace Wellness: Improving Your Experience at Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Ryan Rhodes, Primary investigator, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-108
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Sedentary Behavior; Obesity
MeSH Terms: conditions — Sedentary Behavior; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nutrition condition (Active Comparator): Received nutrition information such as the comparison of nutritional information between orange juice and soda pop. Received intervention following measurements at baseline, week 4, and week 8.
  Interventions: Behavioral: Nutrition condition
- Affective condition (Experimental): Learned about the affective benefits (e.g., less depression) of reduced office sitting time through taking active breaks. Received intervention following measurements at baseline, week 4, and week 8.
  Interventions: Behavioral: Affective condition
- Instrumental condition (Experimental): Learned about instrumental benefits such as the relationship between sitting and cardiovascular disease and absenteeism at work. Received intervention following measurements at baseline, week 4, and week 8.
  Interventions: Behavioral: Instrumental condition
- Self-regulation condition (Experimental): Learned how to self-monitor their sedentary behavior and active breaks. They also learned how to create prompts/cues (e.g., sticky note reminder), problem solve to overcome barriers, action plan (i.e., specifying when, where, and how to do the behavior), and set goals in order to be less sedentary according to SMART (i.e., specific, measurable, attainable, relevant, time-oriented) principles. Received intervention following measurements at baseline, week 4, and week 8.
  Interventions: Behavioral: Self-regulation condition

INTERVENTIONS:
Behavioral: Nutrition condition — Received nutritional information in in-person PowerPoint presentations.
  Arms: Nutrition condition
Behavioral: Affective condition — Received information about affective benefits of less sitting in the workplace in in-person PowerPoint presentations.
  Arms: Affective condition
Behavioral: Instrumental condition — Received information about instrumental benefits of less sitting in the workplace in in-person PowerPoint presentations.
  Arms: Instrumental condition
Behavioral: Self-regulation condition — Learned how to self-regulate behavior to sit less in the workplace in in-person PowerPoint presentations.
  Arms: Self-regulation condition

SUMMARY:
The primary objective of study was to compare affective (i.e., highlighted emotional benefits), instrumental (i.e., highlighted other health benefits), and self-regulation (i.e., demonstrated ways to plan, set goals, etc.) interventions in terms of their ability to motivate less sitting in the workplace. Research of this type is important because people sit for long periods of time at work which adversely affects their health and productivity.

It was hypothesized that the affective and self-regulation groups would sit less than the instrumental and control groups based on evidence indicating that affective attitude (i.e., emotional evaluation of the behavior) and self-regulation techniques tend to predict behavior.

ELIGIBILITY:
Inclusion Criteria:

* From a local workplace in Victoria
* Full-time employee (i.e., greater than 35 hours per week)
* Reported over 5.5 hours of sitting per day at work
* Agreed to attend the 3 intervention sessions

Exclusion Criteria:

* Not from a local workplace in Victoria
* Not a full-time employee (i.e., 35 hours or less per week)
* Reported less than 5.5 hours of sitting per day at work
* Did not agree to attend the 3 intervention sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Sitting time | Twelve weeks post-baseline
  Average hours of sitting time per day at work

CONTACTS AND LOCATIONS:
Locations (1):
- Behavioural Medicine Laboratory, Victoria, British Columbia, Canada

REFERENCES:
- [Derived] Lithopoulos A, Kaushal N, Beauchamp MR, Conner M, de Bruijn GJ, Latimer-Cheung AE, Rhodes RE. Changing Sedentary Behavior in the Office: A Randomised Controlled Trial Comparing the Effect of Affective, Instrumental, and Self-Regulatory Messaging on Sitting. Appl Psychol Health Well Being. 2020 Nov;12(3):687-702. doi: 10.1111/aphw.12202. Epub 2020 May 19. PMID 32428341